CLINICAL TRIAL: NCT01952743
Title: Concomitant Renal Denervation Therapy in Hypertensive Patients Undergoing Atrial Fibrillation Ablation - A Feasibility Study
Brief Title: Renal Denervation Therapy in Hypertensive Patients Undergoing A-Fib Ablation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of efficacy with renal denervation in multicenter trials
Sponsor: Siva Mulpuru (Other)
Responsible Party: Sponsor-Investigator, Siva Mulpuru, M.D., Assistant Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 12-009062
Record Dates: First submitted 2013-09-23; First posted 2013-09-30 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation; Hypertension
Keywords: Atrial Fibrillation; Hypertension; Renal Denervation
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF Ablation alone (Active Comparator): Clinical AF ablation performed as deemed appropriate by operator
  Interventions: Procedure: AF ablation alone
- AF ablation with Renal Denervation (Experimental): Renal denervation performed using the same ablation catheter after clinical AF ablation
  Interventions: Procedure: AF ablation with Renal Denervation

INTERVENTIONS:
Procedure: AF ablation with Renal Denervation — Pulmonary vein isolation (PVI) is performed as per operator preference by previously described techniques. Both mapping and ablation are performed under general anesthesia. The use of standard electrophysiology ablation catheter to perform renal artery ablation in hypertensive patients has been previously described. UP to 2 minutes of RF energy (10W with irrigation flow of 17 ml/min) are delivered at each location and up to 6 lesions for each artery on the longitudinal and rotational axis. Renal denervation is performed on both vascular pedicles after clinical AF ablation in patients assigned to the intervention arm.
  Arms: AF ablation with Renal Denervation
Procedure: AF ablation alone — Pulmonary vein isolation (PVI) is performed as per operator preference by previously described techniques.
  Arms: AF Ablation alone

SUMMARY:
We propose a pilot study to assess safety and benefit of renal artery ablation at the time of planned atrial fibrillation ablation.

DETAILED DESCRIPTION:
Symptomatic atrial fibrillation (AF) refractory to anti-arrhythmic drugs is commonly treated with ablation therapy. Pulmonary vein isolation along with additional substrate medication is commonly performed during ablation procedures is associated with 60-80% success rate for maintenance of sinus rhythm. After AF ablation hypertension (HTN) is a strong predictor for recurrence of atrial fibrillation. Drug resistant hypertension can be effectively treated with catheter based renal denervation therapy. Our primary hypothesis is concomitant renal denervation therapy along with AF ablation is associated with improvement in success rates of AF ablation along with adequate control of blood pressure. The specific objectives of this study are to prospectively compare success rates, time to AF recurrence, AF burden and blood pressure controls in patients randomized to concomitant renal denervation arm when compared to patients with AF ablation alone.

ELIGIBILITY:
Inclusion Criteria:

1. Paroxysmal and Persistent Atrial Fibrillation refractory eligible for AF ablation as per HRS/ECAS/EHRA consensus statement.[23] Paroxysmal AF is defined as two or more episodes of AF lasting less than 7 days in duration during the last 6 months before enrollment. Persistent AF is defined as AF lasting more than 7 days or requiring cardioversion for termination.
2. Hypertension (>140/80 mm Hg) on treatment with at least 1 hypertensive medication.
3. GFR >60ml/dl using Cockcroft- Gault equation

Exclusion Criteria:

1. Secondary causes of hypertension
2. Severe renal artery stenosis or dual renal arteries
3. Congestive heart failure with NYHA class III or IV status
4. EF< 35%
5. LA Diameter >6 cm
6. Previous AF ablation
7. Previous renal artery stent or angioplasty
8. Severe contrast allergy
9. Inability to give informed consent
10. Solitary kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation (AF) Time to recurrence and Burden | 1 year
  After 3 months of blanking period, time to recurrence of atrial arrhythmia lasting more than 30 seconds is measured during follow up. (Atrial fibrillation)AF burden is assessed on a 7 day duration event monitor. Electrocardiogram (EKG) or Event monitor strips will be evaluated by independent board certified physicians.
Hypertension control | 1 year
  BP is obtained as per Joint National Committee (JNC 7) standards at 3, 6 and 12 month visits of follow up. Information regarding titration of antihypertensives or reduction in the number of medications to adequately control blood pressure is collected.

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) at 3, 6 and 12 months | 1 year
Renal artery complications by Crosssectional Imaging (Magnetic Resonance Imaging or computed tomography | 3months
Quality of life scores (MAFSI- Mayo Atrial Fibrillation Symptom Index) | 1 year
Change in left atrial volume parameters | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Siva K. Mulpuru, M.D., Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States